CLINICAL TRIAL: NCT03981445
Title: A Multi-site Multi-Setting Randomized Controlled Trial (RCT) of Integrated HIV Prevention and HCV Care for People Who Inject Drugs (PWID)
Brief Title: Integrated HIV Prevention and HCV Care for PWID
Acronym: M2HepPrEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Université de Montréal (Other); University of Miami (Other); Weill Medical College of Cornell University (Other); Université de Sherbrooke (Other); Simon Fraser University (Other); National Institute on Drug Abuse (NIDA) (NIH); Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Lisa Metsch, Dean of General Studies, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAR5478; R01DA045713 (NIH)
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: HIV Prevention; HCV; Opioid Use; Intravenous Drug Usage
Keywords: PrEP; HCV Treatment; Injection Drug Use

STUDY DESIGN:
Intervention Model Description: This trial is an open-label, multi-site, multi-center, randomized, controlled,superiority trial with two parallel treatment arms. The study is a type-1 hybrid effectiveness implementation study. Participants will be randomized to the on-site integrated care with adherence counselling treatment or the off-site referral to specialized care group with patient navigation in a 1:1 ratio using a permuted-block randomization scheme.
Who Masked: Outcomes Assessor
Masking Description: This trial is an open-label, un-blinded study. Given the pragmatic nature of the trial, participants, providers and research staff will not be blinded. Research and clinical staff will be blinded to the randomization procedure to prevent predictions about participant assignment.Research and clinical staff will initially be blinded to arm assignment to avoid bias, but after baseline the research and clinical staff will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- On-site Integrated Care with Adherence Counseling (Experimental): Participants randomized to the on-site integrated care with adherence counselling arm will be prescribed pre-exposure prophylaxis (PrEP) (Truvada®) and, if indicated, Hepatitis C (HCV) treatment (Epclusa®) at the OAT clinic or SAP from which they were recruited. In addition to PrEP and, if indicated, HCV care, participants in the on-site integrated care arm will receive any required health care services as per local standard of care. Addiction treatment, OAT, and mental health services will be provided, if necessary and available. Participants recruited at syringe access programs (SAP) will be offered addiction counseling and treatment, including OAT when in the integrated care arm in addition to site standard of care.
  Interventions: Behavioral: Adherence Counseling
- Off-site Referral to Specialized Care with Patient Navigation (Experimental): Participants randomized to the off-site referral to specialized care and patient navigation group will be linked to primary care for PrEP and, if necessary, HCV treatment by a patient navigator. Given the replicated success of the AntiRetroviral Treatment Access Study (ARTAS) intervention regarding linking HIV-infected individuals to HIV primary care, we adapted ARTAS to facilitate people who inject drugs linkage with PrEP and, if necessary, HCV treatment services. Participants in the off-site care arm will be prescribed PrEP and, if necessary, HCV treatment by their off-site physician. All necessary care will also be provided to participants by their off-site physician. Off-site physicians will be notified that if their patients are placed on a waiting list, unable to afford, or are otherwise unable to immediately access PrEP or HCV treatment, Truvada® and Epclusa® are available to participants of the M2HepPrEP study immediately and free of charge.
  Interventions: Behavioral: ARTAS Adapted Patient Navigation

INTERVENTIONS:
Behavioral: ARTAS Adapted Patient Navigation — Patient navigation will provided by trained patient navigators to participants randomized to the off-site referral to specialized care arm. Patient Navigators will actively coordinate and link participants to available clinics and community resources by scheduling appointments, arranging transportation, and assisting the participant with completing any paperwork that a clinic or service agent may require. The intervention will include up to five, 30-45 minute face-to-face meetings between the patient navigator and participant. These meetings will be tailored around each participant's needs. Additionally, the patient navigator assists the participant in identifying and utilizing informal and formal sources of support to move along the PrEP and/or HCV care continuum.The patient navigator will help the participant inform off-site physicians of the trial and of the availability of PrEP and HCV medication, should the physician and patient decide to initiate one or both treatments.
  Arms: Off-site Referral to Specialized Care with Patient Navigation
Behavioral: Adherence Counseling — Counseling for PrEP initiation and adherence and, if necessary, HCV treatment will be provided by the clinical counseling staff of the on-site integrated care arm. Adherence counseling will include, but not be limited to, the indications, advantages, and disadvantages (e.g. side effects) of PrEP and HCV treatment in order to help the participant with his/her decision. The counselor will provide any necessary information to the participants and help them to address health and social needs. If required, the counselor will help the patient and physician with insurance-related issues. Adherence counselling will be carried out in a motivational style. The intervention will include five 30-45 minute face-to-face meetings with the participant and the adherence counselor over 6 months.
  Arms: On-site Integrated Care with Adherence Counseling

SUMMARY:
The objective of this study is to compare and evaluate two strategies of delivering PrEP and Hepatitis C Virus (HCV) treatment to people who inject drugs to determine the best method of providing care. Participants will be randomized to one of two treatment arms: on-site integrated care or off-site referral to specialized care.

DETAILED DESCRIPTION:
The first strategy, the on-site integrated care model, provides opioid agonist therapy (OAT) clinics and harm reduction sites/syringe access programs (SAP) with the tools to offer HIV prevention and HCV treatment on-site. The second strategy, the off-site referrals to specialized care model, connects people who are at risk for contracting HIV with patient navigators who help them access available HIV prevention care and, if necessary, HCV treatment.

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet the following criteria to be eligible to participate in the RCT:

1. be 18-64 years of age
2. report injection drug use in the past 6-months
3. be HIV negative
4. provide informed consent
5. complete a medical release form
6. report living in the vicinity and being able to return for follow-up over 18-months
7. be willing to use a medically acceptable form of contraception throughout the study duration (for women of childbearing potential)
8. be able to communicate in English or French (site dependent)
9. be receiving services at an opioid agonist therapy clinic or a syringe access program

Individuals must meet the following criteria to be eligible to participate in the qualitative interview:

1. have completed the first 6 months of RCT follow up (RCT participant interviews);
2. provide informed consent;
3. have contributed to assessments/interviews, intervention and/or treatment follow-ups (staff interviews).

Exclusion Criteria:

Individuals will be excluded from the RCT if they:

1. have any disabling medical conditions as assessed by medical history, physical exam, vital signs, and/or laboratory assessments that in the opinion of the study physician preclude safe participation in the study or ability to provide fully informed consent.
2. have any disabling mental conditions as assessed by medical history and clinical assessment that in the opinion of the study physician precludes safe participation in the study or ability to provide fully informed consent.
3. have chronic renal failure
4. have or have history of decompensated cirrhosis
5. are HIV-positive or have symptoms of an acute HIV infection
6. are pregnant (verified via pregnancy test), are planning to be pregnant during the course of the study, or breastfeeding
7. have an allergy or contraindication to one of the study medications
8. have prior HCV treatment failure with direct-acting antiviral (DAA) regimens (Except those who were treated, cured the virus, but were re-infected with a new virus)
9. are currently on PrEP and/or HCV treatment.
10. are currently in prison, in any inpatient overnight facility as required by court of law or have a pending legal action, which may prevent an individual from completing the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 446 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sustained PrEP adherence | 6 months post randomization
  Average proportion of Dried Blood Spots (DBS) with detectable levels of Tenofovir at 6 months
HCV cure among HCV positive strata | 6-months post treatment initiation
  HCV cure among the HCV positive strata will be compared between both treatment arms at 12 months post randomization. HCV cure is defined as initiating HCV treatment within six (6) months of being randomized and achieving sustained viral response 12 weeks (SVR-12) post-treatment completion. HCV treatment initiation will be measured using self-report and by assessing medical/drug dispensation records. SVR-12 will be measured by testing HCV-RNA negative 12 weeks after end of HCV treatment. If a participant initiates treatment within six (6) months of randomization but does not achieve SVR-12, they will not be counted as a success. Likewise, if a participant who is randomized as HCV positive achieves SVR-12 but did not initiate treatment within 6-months of randomization, they will not be counted as a success.

SECONDARY OUTCOMES:
Long-term sustained PrEP Adherence | Up to 12 months
  Proportion of participants who self-report PrEP use and achieve detectable levels of tenofovir as measured by DBS testing at 6 months and 12 months post randomization.
Behavioral disinhibition | Up to 12 months
  Proportion of participants who increase sexual or injection risk behaviors as measured by self- report questionnaires administered at each research visit.
STI or HIV incidence | Up to 12 months
  Sexually Transmitted Infections (STI) incidence will be defined as a positive test result for Neisseria gonorrhoeae, Chlamydia trachomatis, HIV or syphilis in participants who formerly tested negative for the STI(s).
HCV Incidence | Up to 12 months
  HCV status will be determined by HCV-Ab testing, and if positive, HCV-RNA testing. New incidence of HCV will be defined as an HCV-Ab positive test results in participants who were HCV-Ab negative at a previous testing visit and HCV-Ab positive/HCV-RNA positive test results in participants who had previously tested HCV-Ab positive/HCV-RNA negative
PrEP Initiation/Uptake | Up to 12 months
  Proportion of participants who initiate PrEP before 6 months post randomization and between 6 to 12 months post randomization. PrEP initiation will be defined as record of dispensation of the first dose of TDF/FTC to a participant.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R Metsch, Ph.D, Principal Investigator — Columbia University; Julie Bruneau, M.D., Principal Investigator — Université de Montréal; Daniel Feaster, Ph.D, Principal Investigator — University of Miami; Valérie Martel-Laferrière, MD, Principal Investigator — Université de Montréal
Locations (3):
- United States (2):
  - Miami, Miami, Florida
  - Columbia University Irving Medical Center, New York, New York
- Montreal, Montreal, Quebec, Canada

REFERENCES:
- [Background] Martel-Laferriere V, Feaster DJ, Metsch LR, Schackman BR, Loignon C, Nosyk B, Tookes H, Behrends CN, Arruda N, Adigun O, Goyer ME, Kolber MA, Mary JF, Rodriguez AE, Yanez IG, Pan Y, Khemiri R, Gooden L, Sako A, Bruneau J. M2HepPrEP: study protocol for a multi-site multi-setting randomized controlled trial of integrated HIV prevention and HCV care for PWID. Trials. 2022 Apr 23;23(1):341. doi: 10.1186/s13063-022-06085-3. PMID 35461260
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35461260